CLINICAL TRIAL: NCT07200765
Title: Is the Combination of Ganglion Impar Block and Caudal Epidural Steroid Injection Superior to Ganglion Impar Block Alone in Chronic Coccydynia? A Retrospective Study
Brief Title: Efficacy of Combining Caudal Epidural Steroid With Ganglion Impar Block in Chronic Coccydynia
Status: Active, not recruiting | Type: Observational
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Mesut Bakır, Associate Professor, Mersin University
Other Study IDs: MERSINALG-COCCYDYNIA-2025
Record Dates: First submitted 2025-09-23; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Caudal Epidural Block; Coccygodynia; Coccydynia
Keywords: Chronic Coccydynia, Ganglion impar block

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Ganglion Impar Block: This group includes adults with a diagnosis of chronic coccydynia who underwent a ganglion impar block as part of routine clinical care.The ganglion impar block was performed under fluoroscopic guidance using a transsacrococcygeal approach, with lateral and anteroposterior (AP) views obtained. With the loss-of-resistance technique, the needle was advanced along the intervertebral disc and the ventral tip was positioned anterior to the sacrococcygeal ligament. Needle placement was confirmed by injecting 1 mL of iohexol 350 mg/mL contrast (Omnipaque 350, GE Healthcare, Ireland) into the retroperitoneal space. A total of 5 mL was then administered, consisting of 1 mL methylprednisolone acetate (40 mg/mL), 2 mL normal saline, and 2 mL 0.5% bupivacaine hydrochloride. Outcomes were abstracted from records at baseline, 1 hour, 1 month and 6 month after the procedure.
- Group B: Ganglion Impar Block Combined with Caudal Epidural Steroid Injection: This group includes adults with chronic coccydynia who, as part of routine clinical care, received a combined caudal epidural steroid injection and ganglion impar block. The Caudal Epidural Steroid Injection procedure was performed under fluoroscopic guidance with both lateral and anteroposterior (AP) views. After subcutaneous infiltration of 1 mL of 2% lidocaine, a 22-gauge spinal needle was advanced into the caudal epidural space, and correct placement was confirmed by injection of 1 mL of iohexol 350 mg/mL contrast (Omnipaque 350; GE Healthcare, Ireland). A total of 5 mL was then administered, consisting of 40 mg methylprednisolone acetate diluted in 4 mL of normal saline. Following the caudal epidural steroid injection, the ganglion impar block was performed as described for Group A. Outcomes were abstracted from records at baseline, 1 hour, 1 month and 6 month after the procedure.

SUMMARY:
Coccydynia refers to pain localized to the tailbone (coccygeal) region. Initial management is conservative-nonsteroidal anti-inflammatory drugs (NSAIDs), use of a seat cushion, and physical therapy-yet a proportion of patients remain symptomatic and subsequently pursue interventional options. The ganglion impar block (GIB), originally used to treat perineal cancer pain, is now recognized as an effective approach for perineal and coccygeal pain of both malignant and benign etiologies. Caudal epidural steroid injection (CESI) is also employed, either as monotherapy or in conjunction with other treatments; however, its precise role in coccydynia has not been clearly defined. Evidence directly comparing these injections is limited, and whether the combination confers superiority over GIB alone remains unresolved.

In this retrospective study, we will compare GIB alone versus GIB combined with CESI in adults treated for chronic coccydynia refractory to noninterventional management and evaluate any incremental benefit of the combination.

DETAILED DESCRIPTION:
Coccydynia refers to pain localized to the coccygeal region that commonly intensifies with sitting and forward flexion. It frequently follows a fall or direct trauma and can constrain routine activities. The majority of patients respond to conservative management, including rest, use of a seat cushion, physical therapy, nonsteroidal anti-inflammatory agents, and lifestyle modification. For patients who remain symptomatic, a fluoroscopy-guided ganglion impar block can alleviate pain by modulating sympathetic pathways. The procedure is usually well tolerated; reported complications include infection, bleeding, and, rarely, rectal perforation.

Caudal epidural steroid injection (CESI), administered via the sacral canal, is an adjunctive option used to mitigate inflammation in the lumbosacral region. In selected patients, combining CESI with a ganglion impar block may enhance analgesic control by attenuating inflammation and sympathetic input.

In this retrospective cohort study, the comparative effectiveness of two injection strategies (GIB alone and GIB plus CESI) will be evaluated in adults with chronic coccydynia.

The medical records of patients who presented to the Algology Outpatient Clinic of Mersin University Faculty of Medicine Hospital between January 1, 2020, and May 20, 2025, with chronic coccydynia and who underwent a ganglion impar block will be evaluated in a retrospective review. A minimum target sample size of 50 patients is planned. All included patients had previously received conservative treatment without clinical benefit. Patients were excluded if, at the time of injection, they had an active infection; a history of lumbar or coccygeal surgery; a documented hypersensitivity to local anesthetics or iodinated contrast agents; or a bleeding diathesis. Data collected: age, sex, trauma history, NRS-11 scores pre-procedure, 1 hour, 1 month and 6 month post-procedure.

The ganglion impar block was performed under fluoroscopic guidance using a transsacrococcygeal approach. The injectate volume was 5 mL, consisting of 1 mL methylprednisolone acetate (40 mg/mL), 2 mL normal saline, and 2 mL 0.5% bupivacaine hydrochloride.

The caudal epidural steroid injection (CESI) was performed under fluoroscopic guidance with both lateral and anteroposterior views. A total of 5 mL was administered, comprising 40 mg methylprednisolone acetate diluted in 4 mL normal saline.

Outcome measures included:

Primary: Pain relief measured using a Numerical Rating Scale (NRS) at baseline and 6 months post-procedure.

Secondary: Change in NRS-11 pain score from baseline to 1 hour after the procedure and treatment success rate at 6 months, defined as the proportion of participants achieving ≥50% reduction in NRS-11 pain score or a ≥4-point decrease from baseline (per IMMPACT).

Data was extracted from electronic records and procedure reports. Statistical comparisons will be made using appropriate parametric or non-parametric tests based on data distribution. This study seeks to contribute real-world evidence to guide clinicians in selecting safer, more effective injection strategies for managing chronic coccydynia

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Chronic coccydynia >3 months
* Inadequate response to conservative treatments
* Written informed consent documented for the procedure (per records)

Exclusion Criteria:

* Active infection on the injection date.
* History of lumbar or coccygeal surgery
* Allergy to local anesthetics or contrast media
* Coagulopathy / anticoagulant therapy contraindicating the procedure
* Inadequate follow-up documentation
* Injection performed to a different region during the indexed procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consisted of adults with chronic coccydynia who received either a ganglion impar block (GIB) alone or a combined with caudal epidural steroid injection as part of routine clinical care at the Algology Clinic of Mersin University Hospital between January 1, 2020, and May 20, 2025. Patients were not assigned to treatments by protocol; intervention choice reflected clinician judgment and patient characteristics. Outcomes (e.g., NRS-11 pain scores) were abstracted from medical records at baseline and follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in NRS-11 pain score from baseline to 6 months | Baseline and 6 months post-procedure
  Within-participant change in pain intensity (ΔNRS = 6-month NRS-11 minus baseline NRS-11); negative values indicate improvement. NRS-11: 0=no pain, 10=worst pain.

SECONDARY OUTCOMES:
Treatment success rate at 6 months (IMMPACT) | Baseline and 6 months post-procedure
  Proportion of participants achieving ≥50% reduction in NRS-11 pain score or a ≥4-point decrease from baseline at 6 months (per IMMPACT). Non-responders are all others. NRS-11: 0=no pain, 10=worst pain.
Change in NRS-11 pain score from baseline to 1 hour | Baseline and 1 hour post-procedure.
  Within-participant change in pain intensity (ΔNRS = 1-hour NRS-11 minus baseline NRS-11); negative values indicate improvement. NRS-11: 0=no pain, 10=worst pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Mersin University Faculty of Medicine, Department of Algology, Mersin, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) related to primary and secondary outcomes will be shared upon reasonable request. Data will be available after publication and can be requested by contacting the principal investigator.
Supporting Information: Study Protocol, SAP
Time Frame: De-identified individual participant data and selected supporting documents will be available upon request beginning 6 months after publication. Data will remain available for 5 years.
Access Criteria: Researchers affiliated with academic institutions may request access to anonymized individual participant data and related documents for non-commercial research. Requests must include a brief study proposal and will be reviewed by the principal investigator. Data will be shared via institutional email upon approval.